CLINICAL TRIAL: NCT01066182
Title: A Randomised Controlled Trial of DHA (Docosahexaenoic Acid)for Learning and Behaviour in Children Aged 7 - 9 Years
Brief Title: The DHA (Docosahexaenoic Acid) Oxford Learning and Behaviour (DOLAB) Study
Acronym: DOLAB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Dr. Paul Montgomery, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08/H0603/49; R10157/CN001
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2010-02

CONDITIONS: Learning; Behaviour
Keywords: DHA; Learning; Reading; Memory; Children; Omega 3; Education; Learning and behaviour in children
MeSH Terms: conditions — Behavior | interventions — Docosahexaenoic Acids; Sunflower Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHA supplement (Experimental): 3 x 500 mg capsules per day orally, each capsule providing 200 mg of DHA as a triglyceride. The liquid fill contains DHASCO®-S oil, derived from the microalgae, Schizochytrium sp., high-oleic sunflower oil, natural mixed tocopherols, ascorbyl palmitate, and rosemary extract (flavouring). The gelatin shell contains glycerin, water, and colouring (carmel, carmine, turmeric).
  Interventions: Dietary Supplement: DHA (docosahexaenoic acid)
- Sunflower oil capsule (Placebo Comparator): The placebo will consist of 3 x 500 mg capsules per day orally containing high-oleic sunflower oil. The dimensions, taste, appearance and colour will be identical to those of the DHA capsules. The shell of the capsule will be the same as the DHA capsule. The liquid fill contains high-oleic sunflower oil, natural mixed tocopherols, ascorbyl palmitat and rosemary extract (flavouring).
  Interventions: Dietary Supplement: Sunflower oil capsules

INTERVENTIONS:
Dietary Supplement: DHA (docosahexaenoic acid) — 3 x 500 mg capsules per day orally, each capsule providing 200 mg of DHA as a triglyceride. The liquid fill contains DHASCO®-S oil, derived from the microalgae, Schizochytrium sp., high-oleic sunflower oil, natural mixed tocopherols, ascorbyl palmitate, and rosemary extract (flavouring). The gelatin shell contains glycerin, water, and colouring (carmel, carmine, turmeric).
  Arms: DHA supplement
Dietary Supplement: Sunflower oil capsules — The placebo will consist of 3 x 500 mg capsules per day orally containing high-oleic sunflower oil. The dimensions, taste, appearance and colour will be identical to those of the DHA capsules. The shell of the capsule will be the same as the DHA capsule. The liquid fill contains high-oleic sunflower oil, natural mixed tocopherols, ascorbyl palmitat and rosemary extract (flavouring).
  Arms: Sunflower oil capsule

SUMMARY:
The purpose of this study is to determine whether DHA (in a daily dose of 600 mg.) will improve the behaviour and learning of normal children aged 7-9 years in mainstream state schools who are underperforming according to nationally standardized tests.

DETAILED DESCRIPTION:
The study has two stages, as its primary aim is to find out whether there is a real link between children's fatty acid status and their reading and behaviour. Previous reviews have stated the importance of objective measures, as did our referees.

We will aim to address this by using well validated tests of reading and behaviour, and comparing results from these with children's fatty acid status as assessed from a pinprick blood sample. In Stage 1 we will primarily aim to establish the degree of association between fatty acid status and reading and behaviour. Secondarily, we will look at whether the children who have a higher DHA status have better sleep, and whether in turn they have better reading and/or behaviour, as previous work has suggested this.

In Stage 2 we aim to carry out a randomised trial where children will be given either DHA or a taste- and appearance-matched dummy capsule for 16 weeks. Neither the children, parents nor the researchers will know which children will get which treatment until the study is over.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 7 - 9 years from mainstream state schools who are underperforming in literacy skills according to nationally standardized assessments of scholastic achievement at age 7 years (Key Stage 1 ). To be eligible, children must score below the 33rd centile for reading/writing, but within the normal range in at least one other domain.
2. English as a first language.

Exclusion Criteria:

1. Major learning disabilities or medical disorders
2. Taking medications expected to affect behaviour and learning
3. Taking fish oils already, or eating fish 2 times or more a week

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Conners Teacher Rating Scale (CTRS-L) | 16 weeks
Conners Parent Rating Scale (CPRS-L) | 16 weeks
British Ability Scale (BAS) II Word and Digit Span Scales | 16 weeks

SECONDARY OUTCOMES:
Pinprick blood levels of DHA | 16 weeks
Child Sleep Habits Questionnaire (CSHQ) | 16 weeks
Objective sleep as measured by actigraphy | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Montgomery, DPhil, Principal Investigator — University of Oxford; Alexandra J Richardson, DPhil, Principal Investigator — University of Oxford
Locations (1):
- Department of Social Policy and Social Work, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Richardson AJ, Burton JR, Sewell RP, Spreckelsen TF, Montgomery P. Docosahexaenoic acid for reading, cognition and behavior in children aged 7-9 years: a randomized, controlled trial (the DOLAB Study). PLoS One. 2012;7(9):e43909. doi: 10.1371/journal.pone.0043909. Epub 2012 Sep 6. PMID 22970149